CLINICAL TRIAL: NCT00650988
Title: A Pilot Study of Cryotherapy for Barrett's Esophagus With High-Grade Dysplasia and Early Esophageal Cancers
Brief Title: Cryotherapy for Barrett's Esophagus and Early Esophageal Cancers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE5205; Cleveland Clinic IRB 8270 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Barretts Esophagus; Esophageal Cancer
Keywords: Barrett's Esophagus; Cryospray ablation; High Grade Dysplasia; Early Esophageal Cancers; Esophageal Neoplasms; Esophageal Intramucosal Cancer (IMCA); Esophageal Cancer limited to esophageal wall; Barretts esophagus High Grade Dysplasia (HGD)
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Barrett's Esophagus with intramucosal carcinoma (IMCA) (Experimental)
  Interventions: Procedure: Cryospray Ablation
- Barrett's Esophagus with High Grade Dysplasia (HGD) (Experimental)
  Interventions: Procedure: Cryospray Ablation

INTERVENTIONS:
Procedure: Cryospray Ablation — Liquid nitrogen spray with a cryospray catheter through an upper endoscope that enables the direct visualization of mucosal freeze (cryoburn) of the mucosa treated which avoids the need for direct tissue contact. Frozen state is defined as mucosa appearing white. Cryofreeze is preformed in cycles of 10 second sprays with a minimal thaw of 60 seconds each spray. This cycle is repeated 4 times in each area of treatment.

SUMMARY:
This is a single center study to evaluate the efficacy and safety of a new ablation technique involving the spray of liquid nitrogen through a catheter (cryotherapy) via an upper endoscopy (EGD) to ablate Barrett's esophagus with changes of high-grade dysplasia (HGD) or intramucosal cancer (IMCA) and patients with esophageal cancer limited to the esophageal wall, in whom there are no standard treatment options available.

DETAILED DESCRIPTION:
The Cryo-Ablator System is a cryosurgical unit with a liquid nitrogen cooled cryocatheter and accessories to destroy tissue during surgical procedures by applying extreme cold.

Patients will prepare for esophagogastroduodenoscopy (EGD) in the standard fashion using an overnight fast with only clear liquids and required medications allowed up to 2 hours before the procedure. The EGD will be performed using a therapeutic Olympus endoscope. The cryocatheter is passed into the therapeutic channel of the endoscope. Liquid nitrogen is sprayed through the cryocatheter for a duration of 10 seconds as measured by the device integrated timer. This process will be repeated four times in piecemeal fashion such that for any given area treated it will be maintained in a frozen state for a total of 40 seconds. Following circumferential treatment, the process will be repeated again applying the spray to the same section of mucosa for a duration of 20 seconds. Patients will be contacted the following day to assess for any immediate complications.

Patients will repeat treatment every 6 weeks if no evidence of esophageal mucosal injury, until complete ablation of the Barrett's mucosa has been achieved. Follow up period of five years to monitor healing and progression.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Co-morbid conditions such as severe heart, lung, kidney or liver disease.
* Refusal of surgical intervention after a thorough discussion of the highly experimental nature of cryotherapy.

Group 2:

* Patients with inoperable esophageal cancer (adenocarcinoma oe squamous cell CA) with lesions extending beyond the mucosa but limited to the esophageal wall

Exclusion Criteria:

* Age less than 18 years
* Co-morbid illness expected to cause death within 6 months
* Pregnancy
* Refusal or inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of patients that achieved successful ablation of dysplasia and neoplasia Barrett's Esophagus. | at 12 months from start of treatment
  Determined by the end of protocol biopsies: incremental (absence of HGD and IMCA in all specimens); partial (residual IMCA with absence of any dysplasia); complete (absence of any intestinal metaplasia or dysplasia)
Number of patients that experience toxicity with cryotherapy | at 12 months from start of therapy
  Toxicity is defined as death or esophageal perforation

SECONDARY OUTCOMES:
Assess the degree of tumor ablation of inoperable early esophageal cancer | at 12 months from start of therapy
  Number of patient with each response determined by the end of protocol biopsies: incremental (absence of HGD and IMCA in all specimens); partial (residual IMCA with absence of any dysplasia); complete (absence of any intestinal metaplasia or dysplasia); no response

CONTACTS AND LOCATIONS:
Overall Officials: John A. Dumot, D.O., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States